CLINICAL TRIAL: NCT07001761
Title: Ultrasonographic Evaluation of Osteoarthritis. A Comparative Study to Conventional Radiography in Patients With Painful Knee.
Brief Title: Ultrasonographic Evaluation of Osteoarthritis.
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Mohamed Elaref, Resident doctor at radiology department Sohag University, Sohag University
Other Study IDs: Noha Mohamed Elaref
Record Dates: First submitted 2025-05-21; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — High-Energy Shock Waves; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Ultrasound/ x rays — * The MSK Ultrasound (US) will be performed using a General Electric LOGIQ P9 unit / Toshiba Applio 500 unit using a 7-13 MHz linear array transducer.
  * Conventional Radio-graphic examination bi-plane weight-bearing semi-flexed (15) radiograms will be taken of the target knee; one in the posteroanterior view, and one in the lateral medial view

SUMMARY:
Assessment of the effectiveness of ultrasonography in correlation to conventional imaging for the detection of the definite grading of knee osteoarthritis.

DETAILED DESCRIPTION:
Assessment the effectiveness of ultrasonography in correlation to conventional imaging for the detection of the definite grading and the complication of knee osteoarthritis for patient complaining from knee pain coming to our radiology department for imaging with a clinical signs of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

Age: above 30 years. Unilateral or bilateral knee joint affection. Symptomatic patient.

Exclusion Criteria:

* Any female patient in the child bearing period presented with Chronic inflammatory joint disease as Rheumatoid arthritis, SLE. Systemic diseases: Renal failure. Significant joint trauma or surgery.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
The outcome for the study is to test the MUS score's ability to discern various degrees of knee OA, in comparison with plain radiography and the 'Knee injury and Osteoarthritis Outcome Score' (KOOS). | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt